CLINICAL TRIAL: NCT03623477
Title: Can Cognitive Training Decrease Reactive Aggression? The Role of Improved Emotion Regulation, Emotion Awareness, and Impulse Control
Brief Title: Can Cognitive Training Decrease Reactive Aggression?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Brain & Behavior Research Foundation (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1505016194; UL1TR000457 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2018-08-09 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Schizophrenia; Cognitive Deficits; Impulsive Aggression; Emotion; Impulsivity
Keywords: Cognitive Remediation; Social Cognition Training; Emotion Regulation; Urgency
MeSH Terms: conditions — Schizophrenia; Cognition Disorders; Impulsive Behavior; Emotional Regulation | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Remediation (CRT) (Active Comparator): Participants assigned to CRT alone will complete 24 hours of neurocognitive training activities and 12 hours of control computer activities.
  Interventions: Behavioral: Cognitive Remediation (CRT)
- CRT+ Social Cognition Training (Experimental): Participants assigned to the combination of CRT and SCT will complete 24 hours of computerized neurocognitive training in memory, attention, and processing speed, and 12 hours of computerized social cognition training focused on improving emotion recognition, social perspective taking, and mentalizing abilities.
  Interventions: Behavioral: CRT+ Social Cognition Training

INTERVENTIONS:
Behavioral: Cognitive Remediation (CRT) — Study compares two configurations of cognitive training--computerized cognitive remediation versus a combination of computerized cognitive remediation and social cognition training. The cognitive remediation therapy group will complete computerized training activities in attention, memory, processing speed, problem solving, and executive functions.
  Arms: Cognitive Remediation (CRT)
Behavioral: CRT+ Social Cognition Training — Study compares two configurations of cognitive training--computerized cognitive remediation versus a combination of computerized cognitive remediation and social cognition training. The combined cognitive remediation and social cognition training group will complete computerized training that target neurocognitive functions, facial affect emotion recognition and mentalizing tasks.
  Arms: CRT+ Social Cognition Training

SUMMARY:
The purpose of the study is to examine the effects of cognitive training on emotion regulation, impulse control, and aggression in people with schizophrenia. The study compares a combination of computerized cognitive remediation and social cognition training (CRT+SCT) to cognitive remediation alone (CRT). Study outcomes include multiple measures of aggression, emotion regulation, impulse control, cognition, and symptoms.

DETAILED DESCRIPTION:
Neurocognitive and social cognitive impairments are contributors to negative emotionality and impulsive aggression in people with schizophrenia. Impulsive aggression poses several challenges to the care of people with schizophrenia. These include a greater risk of rehospitalization and longer hospital stays, involvement with the criminal justice system, and increased risk of recidivism. The investigators recently found that schizophrenia patients with aggression history experienced improvements in neurocognition as well as decreased hostility/agitation and incidents of verbal and physical aggression after participating in cognitive remediation training (CRT). Based on these findings, it is hypothesized that improving neurocognition through CRT may have enhanced the capacity of schizophrenia patients to inhibit aggression through improved emotion regulation capacity and impulse control. It is also postulated that the addition of Social Cognition Training (SCT) to CRT would provide greater benefits on emotion regulation and impulse control over CRT alone. To test the hypotheses, the investigators will conduct a clinical trial that compares two configurations of cognitive training--CRT plus SCT versus CRT plus control computer games. The goal of the study is to examine the comparative benefits of the two configurations of cognitive training on outcomes that include neurocognition, social cognition, emotion regulation, impulse control, and reactive aggression. Participants assigned to the CRT plus SCT group will complete 24 hours of CRT and 12 hours of SCT. Participants assigned to the CRT only group will complete 24 hours of CRT and 12 hours of control computer activities. Emotion regulation, impulse control, and reactive aggression will be indexed using laboratory-based challenges. The investigators will recruit and characterize 90 study participants on demographic and clinical variables including age, gender, education, aggression history, and medications. Study outcome measures will be administered at baseline and posttreatment to participants randomized to the study groups. In a subsample of 32 patients, the study investigators will further examine changes in the neural network of emotion regulation and impulsivity before and after cognitive training.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizo-affective disorder
* Age 18-60
* Mini Mental Status Exam score greater/equal to 24 at screening
* Auditory and visual acuity adequate to complete cognitive tests
* At least a score of 5 or more on the Life History of Aggression (LHA) aggression items or one confirmed assault in the past year
* Capacity and willingness to give consent

Exclusion Criteria:

* Inability to read or speak English
* Documented significant disease of the Central Nervous System (CNS)
* History of intellectual impairment predating psychosis (e.g., a diagnosis of developmental disability)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Aggression | Change from baseline in aggression measures up to the end of intervention at 4 months
  Overt Aggression Scale-Modified (OAS-M); Taylor Aggression Paradigm (TAP); Point Subtraction Aggression Paradigm (PSAP).

SECONDARY OUTCOMES:
Change in cognitive outcomes | Change from baseline in cognition measures up to the end of intervention at 4 months
  MATRICS Consensus Cognitive Battery (MCCB); Emotion Recognition-40 (ER-40); Reading the Mind in the Eyes (Eyes Task)
Change in Emotionality | Change from baseline in emotionality measures up to the end of intervention at 4 months
  Positive and Negative Affect Scale (PANAS); Toronto Alexithymia Scale (TAS); Observer Alexithymia Scale (OAS)
Change in Emotion Regulation Capacity | Change from baseline in measures up to the end of intervention at 4 months
  Picture viewing task completed while peripheral psychophysiological response is obtained
Change in Impulse Control | Change from baseline in impulse control measures up to the end of intervention at 4 months
  Behavioral Impulse control tasks including Go-NoGo Task and Emotional Stop Task

OTHER OUTCOMES:
Change in psychotic symptoms | Change from baseline in psychotic symptom measure up to the end of intervention at 4 months
  Positive and Negative Syndrome Scale (PANSS). Scale total scores range from 30 to 210 with higher scores indicating greater symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony O Ahmed, PhD, Principal Investigator — Weill Medical College of Cornell University; Jean-Pierre Lindenmayer, MD, Principal Investigator — Manhattan Psychiatric Center; Matthew J Hoptman, PhD, Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (2):
- United States (2):
  - Manhattan Psychiatric Center, New York, New York
  - NewYork Presbyterian Hospital, White Plains, New York

IPD SHARING:
Plan to Share IPD: No